CLINICAL TRIAL: NCT02957474
Title: A Phase 1, Open Label, Single Center, Randomized, Six-Sequence, Crossover Study to Evaluate the Effect of Food, Formulation Strength, and a Proton Pump Inhibitor on GED 0301 Pharmacokinetics in Healthy Adult Subjects
Brief Title: A Study to Evaluate the Effect of Food, Formulation Strength, and a Proton Pump Inhibitor on GED 0301 Pharmacokinetics in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GED-0301-CP-001
Record Dates: First submitted 2016-11-03; First posted 2016-11-07 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2017-01

CONDITIONS: Healthy Volunteers
Keywords: Healthy Volunteers; Pharmacokinetics; Food Effect; Proton Pump; GED-0301; Mongersen
MeSH Terms: interventions — GED0301; Omeprazole

ARMS (4):
- Treatment A = single oral dose GED 0301, fasted (Experimental): Subjects will receive a single oral 160 mg dose of GED-0301 after a 10 hour overnight fast
  Interventions: Drug: GED-0301
- Treatment B = single oral dose GED 0301, fed (Experimental): Subjects will receive a single oral 160 mg dose of GED-0301 after a 10 hour overnight fast, and within 30 minutes of completely consuming a high fat meal.
  Interventions: Drug: GED-0301
- Treatment C = single oral dose GED 0301 fasted (Experimental): Subjects will receive an oral dose of 160 mg of GED-0301 given as 4 tablets of 40 mg, after a 10 hour overnight fast
  Interventions: Drug: GED-0301
- Treatment D = oral omeprazole and GED-0301 (Experimental): Subjects will receive one oral dose of 40 mg omeprazole once a day for 6 days. On the 5th day, a single oral 160 mg dose of GED-0301 will be given together with omeprazole.
  Interventions: Drug: GED-0301; Drug: Omeprazole

INTERVENTIONS:
Drug: GED-0301
  Other Names: Mongersen
Drug: Omeprazole
  Arms: Treatment D = oral omeprazole and GED-0301

SUMMARY:
This is an open label, single-center, 4-period, 6-sequence study in healthy subjects to compare the PK of GED 0301 after a single oral dose in the fed and fasted state, and after co administration with omeprazole, a proton pump inhibitor.

The study will consist of a screening phase, a baseline phase, four treatment periods, and a follow up phone call five days (± 1 day) after discharge.

DETAILED DESCRIPTION:
Subjects will be consented and screened within 21 days of dosing. They will undergo routine screening procedures including physical examinations (PE), 12 lead electrocardiograms (ECGs), vital sign measurements, clinical laboratory safety tests (clinical chemistry, haematology, urinalysis), pregnancy tests for females, and serology/drug/alcohol screens.

Eligible subjects will return to the clinic site on Day -1 for baseline safety assessments. After an overnight fast of at least 10 hours, subjects will be assigned randomly to one of six treatment sequences which will determine fasting status and the order in which treatments will be administered.

Subjects in the fasted arm will receive either a single 160 mg tablet of GED 0301 or four 40 mg tablets of GED 0301, with approximately 240 mL of room temperature, non-carbonated water.

Subjects in the fed arm will be required to fast overnight for at least 10 hours. On the morning of dosing, these subjects will be served a high-fat meal. The meal should be entirely consumed within 20 minutes of being served. Dosing of a single160 mg tablet of GED 0301 will occur within 30 minutes (± 5 minutes) after the start of the meal.

During the fourth period, subjects will receive once daily oral doses of 40 mg omeprazole for 6 days (Days 10 through 16). Subjects will fast on the evening of the fourth day for at least 10 hours prior to receiving the last treatment, which is a single dose of 160 mg GED 0301 together with one 40 mg oral dose of omeprazole (Day 15). On Day 16, subjects will take the last dose of omeprazole.

Serial blood sampling for the determination of GED 0301 levels in plasma will be performed during each period for 48 hours post dose.

Subjects will be domiciled at the clinic site from Day 1 of Period 1 until Day 17. All subjects will be discharged from the clinic site on Day 17 when all required safety and PK procedures have been completed.

A follow up phone call will occur five days (± 1 day) after discharge from the clinic center.

The study will be conducted in compliance with Good Clinical Practice (GCP), as described in International Conference on Harmonisation (ICH) Guideline E6 and in accordance with the general ethical principles outlined in the Declaration of Helsinki. The study will receive approval from an EC prior to commencement. The Investigator will conduct all aspects of this study in accordance with applicable national, state, and local laws of the pertinent regulatory authorities.

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subject is male, or non-pregnant and non-nursing female ≥ 18 and ≤ 65 years of age the time of signing the ICF.
2. Subject must understand and voluntarily sign an ICF prior to any study related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements.
4. Satisfactory medical assessment with no clinically significant or relevant abnormalities as determined by medical history, physical examination, vital signs, 12-lead ECG, and clinical laboratory evaluation (haematology, biochemistry, coagulation, and urinalysis) that is reasonably likely to interfere with the subject's participation in or ability to complete the study as assessed by the Investigator.
5. Female subjects NOT of childbearing potential must:

   1. Have been surgically sterilized (hysterectomy or bilateral oophorectomy; proper documentation required) at least 6 months before screening, or be postmenopausal (defined as 24 consecutive months without menses before screening, with a follicle stimulating hormone [FSH] level of > 40 IU/L at screening).
6. Females of childbearing potential (FCBP) must have a negative pregnancy test at the Screening and Baseline Visits. While receiving investigational product (IP) and for at least 28 days after taking the last dose of IP, FCBP who engage in activity in which conception is possible must use one of the approved contraceptive options described below:

   Option 1: Any one of the following highly effective methods: hormonal contraception (oral, injection, implant, transdermal patch, vaginal ring); intrauterine device (IUD); tubal ligation; or partner's vasectomy.

   OR Option 2: Male or female condom PLUS 1 additional barrier method: (a) diaphragm with spermicide; (b) cervical cap with spermicide; or (c) contraceptive sponge with spermicide.
7. Male subjects must:

   a. Practice true abstinence (which must be reviewed on a monthly basis and source documented) or agree to use a barrier method of birth control (condoms not made out of natural [animal] membrane [latex condoms are recommended]) during sexual contact with a pregnant female or FCBP while participating in the study, during dose interruptions, and for at least 28 days after the last dose of IP, even if he has undergone a successful vasectomy.
8. Subject has body mass index (BMI) ≥ 18 and ≤ 33 kg/m2 at screening.
9. Subject has clinical laboratory safety test results that are within normal limits or acceptable to the Investigator.
10. Subject vitals are as follows:

    1. Tympanic body temperature: 35.0 - 37.5°C.
    2. Supine blood pressure (BP) after at least 5 minutes supine rest:

    i. Systolic BP: 90 - 140 mmHg ii. Diastolic BP: 40 - 90 mmHg c. Supine heart rate (after at least 5 minutes of rest): 40 - 90 beats per minute d. Postural drop (standing BP taken after no more than 1 minute standing) of ≤20 mmHG (systolic) or ≤10 mmHg (diastolic) associated with clinically relevant symptoms.
11. Subject has a normal or clinically acceptable 12 lead ECG at screening. In addition:

    1. If male, subject has a QTcF value ≤ 430 msec at screening.
    2. If female, subject has a QTcF value ≤ 450 msec at screening.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Subject has any significant and relevant medical condition (including but not limited to neurological, gastrointestinal, renal, hepatic, cardiovascular, psychological, pulmonary, metabolic, endocrine, hematological, allergic disease, drug allergies, or other major disorders), laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Subject has any condition that confounds the ability to interpret data from the study.
4. Subjects who have:

   a. previously been exposed to GED 0301; or b. been exposed to an investigational drug (new chemical entity) within 90 days preceding the first dose administration, or five half-lives of that investigational drug, if known (whichever is longer).
5. Subject has used any prescription drugs or over-the-counter medication (including multi-vitamins) in the 14 days prior to the planned admission day.

1. Subject has consumed herbal remedies or dietary supplements containing St. John's Wort, in the three weeks before the planned admission day.

6. Subject has any surgical or medical conditions possibly affecting drug absorption, distribution, metabolism, and excretion, eg, bariatric procedure. Appendectomy and cholecystectomy are acceptable.

7. Subject donated blood or plasma within 8 weeks before the first dose administration to a blood bank or blood donation center.

8. Subject has a history of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before the first dose administration, or positive drug screening test reflecting consumption of illicit drugs.

9. Subject has a history or clinical evidence of substance and/or alcohol abuse within the 12 months before screening. Alcohol abuse is defined as regular weekly intake of more than 14 units (using alcohol tracker http://www.nhs.uk/Tools/Pages/NHSAlcoholtracker.aspx).

10. Subject is known to have serum hepatitis or known to be a carrier of hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.

11. Subject smokes > 10 cigarettes per day, or the equivalent in other tobacco products (self reported).

12. Subject is part of the clinical staff personnel or a family member of the clinical site staff.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2016-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics - Cmax | Up to Day 17
  Maximum observed concentration in plasma
Pharmacokinetics -AUC0-∞ | Up to Day 17
  Estimation of AUC from time zero extrapolated to infinity

SECONDARY OUTCOMES:
Adverse Event (AE) | Up to Day 22
  Number of participants with adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Maria Palminsano, MD, Study Director — Celgene Corporation
Locations (1):
- Richmond Pharmacology, Ltd., Croydon, Surrey, United Kingdom